CLINICAL TRIAL: NCT02709512
Title: Randomized, Double-Blind, Phase 2/3 Study in Subjects With Malignant Pleural Mesotheliomato Assess ADI-PEG 20 With Pemetrexed and Cisplatin (ATOMIC-Meso Phase 2/3 Study)
Brief Title: Ph 2/3 Study in Subjects With MPM to Assess ADI-PEG 20 With Pemetrexed and Cisplatin
Acronym: ATOMIC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POLARIS2015-003
Record Dates: First submitted 2016-03-05; First posted 2016-03-16 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-08

CONDITIONS: Mesothelioma
Keywords: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — ADI PEG20; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: ADI-PEG 20 plus Pem Platinum (Experimental): Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM) Duration : Course of Study
  In Combination With:
  Pemetrexed Dose: 500 mg/m2 every 3 weeks Route of Administration: Intravenous Cisplatin Dose: 75 mg/m2 every 3 weeks Route of Administration: Intravenous Carboplatin Dose: AUC 5 mg/mL/min every 3 weeks Route of Administration: Intravenous
  ADI-PEG 20 plus Pem Platinum: Investigational Drug in combination approved standard of care treatment for this indication
  Interventions: Drug: ADI-PEG 20 plus Pem Platinum
- Drug: Placebo plus Pem Platinum (Placebo Comparator): Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM) Duration : Course of Study
  In Combination With:
  Pemetrexed Dose: 500 mg/m2 every 3 weeks Route of Administration: Intravenous Cisplatin Dose: 75 mg/m2 every 3 weeks Carboplatin Dose: AUC 5 mg/mL/min every 3 weeks Route of Administration: Intravenous
  Placebo plus Pem Platinum: Placebo in combination approved standard of care treatment for this indication
  Interventions: Other: Placebo plus Pem Platinum

INTERVENTIONS:
Drug: ADI-PEG 20 plus Pem Platinum — Investigational Drug in combination approved standard of care treatment for this indication
  Other Names: Pemetrexed; Cisplatin; Carboplatin
  Arms: Drug: ADI-PEG 20 plus Pem Platinum
Other: Placebo plus Pem Platinum — Placebo in combination approved standard of care treatment for this indication
  Other Names: Pemetrexed; Cisplatin; Carboplatin
  Arms: Drug: Placebo plus Pem Platinum

SUMMARY:
This is a study of ADI-PEG 20 (pegylated arginine deiminase), an arginine degrading enzyme versus placebo in patients with malignant pleural mesothelioma. Malignant pleural mesothelioma have been found to require arginine, an amino acid. Thus the hypothesis is that by restricting arginine with ADI-PEG 20, the malignant pleural mesothelioma cells will starve and die.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven unresectable MPM of biphasic or sarcomatoid histology
* Naïve to chemotherapy or immunotherapy
* ECOG PS 0-1
* Expected survival of at least 3 months
* Age 18 years or over (there is no upper age limit)
* Measurable disease by modified RECIST criteria for MPM for local pleural disease and RECIST 1.1 criteria for metastatic lesions
* Written (signed and dated) informed consent and must be capable of co-operating with treatment and follow up
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Radiotherapy (except for palliative reasons) in the previous two weeks before study treatment
* History of unstable cardiac disease
* Ongoing toxic manifestations of previous treatments
* Symptomatic brain or spinal cord metastases (patients must be stable for > 1 month post radiotherapy or surgery)
* Major thoracic or abdominal surgery from which the patient has not yet recovered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Bomalaski, MD, Study Director — Polaris Group
Locations (45):
- United States (10):
  - Mayo Clinic, Phoenix, Arizona
  - UCLA Hematology & Oncology - Santa Monica, Los Angeles, California
  - University of California San Francisco Helen Diller Comprehensive Cancer Center, San Francisco, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University of Maryland, Marlene & Stewart Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Tweed Hospital (NNSW LHD), Tweed Heads, New South Wales
  - Princess Alexandria Hospital and Health Services, Woolloongabba, Queensland
  - Southern Adelaide Local Health Network, Inc., Bedford Park, South Australia
  - Austin Health, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Italy (9):
  - SS. Antonio e Biagio e Cesare Arrigo Hospital, Alessandria, AL
  - Humanitas Gavazzeni, Bergamo, BG
  - Ospedale Villa Scassi, Genova, GE
  - Azienda Ospedaliera San Gerardo - Monza, Chirurgia Toracica, Monza, MB
  - European Institute of Oncology, Milan, MI
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Fondazione IRCCS - Istituto Nazionale dei Tumori Milano, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Foundation LinKou Branch, Taoyuan District
- United Kingdom (14):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Plymouth Hospitals (Derriford Hospital), Plymouth, Devon
  - Centre for Experimental Cancer Medicine (CECM), London, England
  - Southampton General Hospital, Southampton, Hampshire
  - University Hospitals Leicester, Leicester, Leicestershire
  - Scunthorpe General Hospital, Scunthorpe, North Lincolnshire
  - Wansbeck General Hospital, Ashington, Northumberland
  - Oxford Cancer and Haematology Centre, The Churchill Hospital, Oxford, Oxfordshire
  - Velindre Cancer Centre, Cardiff
  - Edinburgh Cancer Centre, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - St Bartholomew's Hospital, London
  - University Hospital of South Manchester, Manchester

REFERENCES:
- [Derived] Szlosarek PW, Creelan BC, Sarkodie T, Nolan L, Taylor P, Olevsky O, Grosso F, Cortinovis D, Chitnis M, Roy A, Gilligan D, Kindler H, Papadatos-Pastos D, Ceresoli GL, Mansfield AS, Tsao A, O'Byrne KJ, Nowak AK, Steele J, Sheaff M, Shiu CF, Kuo CL, Johnston A, Bomalaski J, Zauderer MG, Fennell DA; ATOMIC-Meso Study Group. Pegargiminase Plus First-Line Chemotherapy in Patients With Nonepithelioid Pleural Mesothelioma: The ATOMIC-Meso Randomized Clinical Trial. JAMA Oncol. 2024 Apr 1;10(4):475-483. doi: 10.1001/jamaoncol.2023.6789. PMID 38358753
- [Derived] Szlosarek PW, Phillips MM, Pavlyk I, Steele J, Shamash J, Spicer J, Kumar S, Pacey S, Feng X, Johnston A, Bomalaski J, Moir G, Lau K, Ellis S, Sheaff M. Expansion Phase 1 Study of Pegargiminase Plus Pemetrexed and Cisplatin in Patients With Argininosuccinate Synthetase 1-Deficient Mesothelioma: Safety, Efficacy, and Resistance Mechanisms. JTO Clin Res Rep. 2020 Sep 3;1(4):100093. doi: 10.1016/j.jtocrr.2020.100093. eCollection 2020 Nov. PMID 34589965
- [Derived] Uprety D. CheckMate 743: A Glimmer of Hope for Malignant Pleural Mesothelioma. Clin Lung Cancer. 2021 Mar;22(2):71-73. doi: 10.1016/j.cllc.2020.11.009. Epub 2020 Dec 2. No abstract available. PMID 33358660

RESULTS

PARTICIPANT FLOW:
Period: Phase 2
Arm/Group | Drug: ADI-PEG 20 Plus Pem Platinum | Drug: Placebo Plus Pem Platinum
Started | 87 | 89
Completed | 87 | 89
Not Completed | 0 | 0
Period: Phase 3
Arm/Group | Drug: ADI-PEG 20 Plus Pem Platinum | Drug: Placebo Plus Pem Platinum
Started | 125 | 124
Completed | 125 (For Phase 3 the total number of subjects enrolled included 87 subjects from Phase 2 that counted towards 125 enrolled subjects on this arm.) | 124 (For Phase 3 the total number of subjects enrolled included 89 subjects from Phase 2 that counted towards 124 enrolled subjects on this arm.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: ADI-PEG 20 Plus Pem Platinum | Drug: Placebo Plus Pem Platinum | Total
Number analyzed (Participants) | 125 | 124 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (7.98) | 69.4 (7.91) | 69.4 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 102 | 104 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 119 | 117 | 236
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 116 | 116 | 232
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Objective Response Rate is calculated as the proportion of subjects whose best tumor response from all post-baseline tumor assessments is complete response (CR) or partial response (PR). The best tumor response is the best response recorded from the start of the treatment until the end of treatment taking into account any requirement for confirmation.
  To test Objective Response Rate significance, a Relative Risk Ratio (ADI-PEG 20 / Placebo) was calculated as the common relative risk of having a response (CR or PR) based on the Mantel-Haenszel estimator controlling for tumor histology (biphasic versus sarcomatoid).
Time Frame: approximately 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: ADI-PEG 20 Plus Pem Platinum | Drug: Placebo Plus Pem Platinum
Number analyzed (Participants) | 87 | 89
Participants | 12 | 12
Statistical Analysis 1: Comparison: Drug: ADI-PEG 20 Plus Pem Platinum vs Drug: Placebo Plus Pem Platinum; Test type: Superiority — Relative Risk Ratio (ADIPemPlatinum/PlaceboPemPlatinum) is the common relative risk of having a response (CR or PR) based on the Mantel-Haenszel estimator controlling for tumor histology. A relative risk ratio greater than one is favorable to ADIPemPlatinum; p = 0.9489, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.50 to 2.11]

2. Primary Outcome: Overall Survival Phase 3 Interim Analysis
Description: The primary analysis of OS Phase 3 was performed at the interim analysis. This was performed once 50% of the planned OS events for phase 3 have occurred (ie, 169 of the 338 planned OS events). This interim analysis will evaluate OS in the ITT population in an unblinded manner. The OS data at the second interim analysis will be analyzed to support the following decisions:
  Futility stopping: Terminate the study due to futility at the interim analysis. Sample size re-estimation: Increase the target number of OS events after the second interim analysis.. The treatment effect on OS will be evaluated using the stratified log-rank test (stratified by tumor histology).
Time Frame: Approximately 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Drug: ADI-PEG 20 Plus Pem Platinum | Drug: Placebo Plus Pem Platinum
Number analyzed (Participants) | 78 | 91
months | 9.82 [7.85 to 12.91] | 7.49 [5.88 to 9.46]
Statistical Analysis 1: Comparison: Drug: ADI-PEG 20 Plus Pem Platinum vs Drug: Placebo Plus Pem Platinum; Test type: Superiority; p = 0.0078, Log Rank; Cox Proportional Hazard = 0.64, 95% CI 2-sided [0.47 to 0.88]

3. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death. In the event that no death was documented prior to study termination or analysis cutoff, OS was censored at the last known date the subject was known to be alive, either through completion of on-study visits or through survival follow-up contact.
  The treatment effect on OS was evaluated using the stratified log-rank test (stratified by tumor histology).
  The Kaplan-Meier curves were also plotted. A Cox proportional hazard model with an adjustment for tumor histology (biphasic vs sarcomatoid) was used to compute the estimated hazard ratio and two-sided 95% CI. The treatment effect on OS was evaluated using the stratified log-rank test (stratified by tumor histology). The significance level to be used in the OS analysis at the final analysis was based on α = 0.04999 (two-sided).
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Drug: ADI-PEG 20 Plus Pem Platinum: Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM) Duration : Course of Study
  In Combination With:
  Pemetrexed Dose: 500 mg/m2 every 3 weeks Route of Administration: Intravenous Cisplatin Dose: 75 mg/m2 every 3 weeks Route of Administration: Intravenous Carboplatin Dose: AUC 5 mg/mL/min every 3 weeks Route of Administration: Intravenous
  ADI-PEG 20 plus Pem Platinum: Investigational Drug in combination approved standard of care treatment for this indication
  ADI-PEG 20 plus Pem Platinum: Investigational Drug in combination approved standard of care treatment for this indication
- Drug: Placebo Plus Pem Platinum: Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM) Duration : Course of Study
  In Combination With:
  Pemetrexed Dose: 500 mg/m2 every 3 weeks Route of Administration: Intravenous Cisplatin Dose: 75 mg/m2 every 3 weeks Carboplatin Dose: AUC 5 mg/mL/min every 3 weeks Route of Administration: Intravenous
  Placebo plus Pem Platinum: Placebo in combination approved standard of care treatment for this indication
  Placebo plus Pem Platinum: Placebo in combination approved standard of care treatment for this indication
Arm/Group | Drug: ADI-PEG 20 Plus Pem Platinum | Drug: Placebo Plus Pem Platinum
Number analyzed (Participants) | 108 | 116
months | 9.30 [7.85 to 11.79] | 7.66 [6.14 to 9.53]
Statistical Analysis 1: Comparison: Drug: ADI-PEG 20 Plus Pem Platinum vs Drug: Placebo Plus Pem Platinum; Test type: Superiority; p = 0.0234, Log Rank; Cox Proportional Hazard = 0.71, 95% CI 2-sided [0.55 to 0.93]

4. Secondary Outcome: Progression Free Survival
Description: The key secondary endpoint for the phase 3 portion is PFS, which will be analyzed only if the analysis of OS is statistically significant at the final analysis, with alpha level of 0.05 (two-sided) using the same statistical methodologies as applied to OS.
Time Frame: approximately 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Drug: ADI-PEG 20 Plus Pem Platinum | Drug: Placebo Plus Pem Platinum
Number analyzed (Participants) | 74 | 71
months | 6.24 [5.78 to 7.43] | 5.65 [4.14 to 5.91]
Statistical Analysis 1: Comparison: Drug: ADI-PEG 20 Plus Pem Platinum vs Drug: Placebo Plus Pem Platinum; Test type: Superiority; p = 0.0193, Log Rank; Cox Proportional Hazard = 0.65, 95% CI 2-sided [0.46 to 0.90]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected with onset after the first dose of study drug or existing events that worsened after the first dose during the study, approximately 18 months.
Arm/Group | Drug: ADI-PEG 20 Plus Pem Platinum | Drug: Placebo Plus Pem Platinum
All-Cause Mortality (participants affected / at risk) | 62/125 | 61/124
Serious Adverse Events (participants affected / at risk) | 19/125 | 20/124
Other Adverse Events (participants affected / at risk) | 106/125 | 111/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: ADI-PEG 20 Plus Pem Platinum (N=125) | Drug: Placebo Plus Pem Platinum (N=124)
Pneumonia (Infections and infestations) | 5 (19) | 6 (20)
Pyrexia (General disorders) | 5 (15) | 8 (11)
Nausea (Gastrointestinal disorders) | 1 (9) | 7 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 2 (7)
Atrial Fibrillation (Cardiac disorders) | 4 (9) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 6 (6) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Musculoskeletal Testing (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (7)
Cerebrovascular Accident (Nervous system disorders) | 1 (3) | 3 (6)
Fall (Injury, poisoning and procedural complications) | 2 (5) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (4)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Anaphylactic Reaction (Immune system disorders) | 2 (4) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (19) | 6 (20)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: ADI-PEG 20 Plus Pem Platinum (N=125) | Drug: Placebo Plus Pem Platinum (N=124)
Nausea (Gastrointestinal disorders) | 65 (106) | 67 (111)
Fatigue (General disorders) | 66 (106) | 62 (111)
Constipation (Gastrointestinal disorders) | 54 (106) | 41 (111)
Anemia (Blood and lymphatic system disorders) | 34 (106) | 38 (111)
Decreased Appetite (Metabolism and nutrition disorders) | 26 (106) | 44 (111)

LIMITATIONS AND CAVEATS:
Enrollment stopped early at the recommendation of the DSMB due to interim analysis positive results and because of slow study enrollment related to an evolving treatment landscape for MPM and the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT02709512/Prot_SAP_000.pdf